CLINICAL TRIAL: NCT03472911
Title: Minimum Effective Volume of Bupivacaine 0.5% for Ultrasound-guided Retroclavicular Approach to Infraclavicular Brachial Plexus Block
Brief Title: Retroclavicular Approach to Infraclavicular Block
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: AntalyaTRH 20
Record Dates: First submitted 2018-03-15; First posted 2018-03-21 (Actual); Last update posted 2018-05-03 (Actual); Status verified 2018-01

CONDITIONS: Bupivacaine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: minimum effective volume — The determination of MEV50 and its 95% confidence interval (CI) was based on the staircase up-and-down method by Dixon and Massey.

SUMMARY:
In this study, the primary objective was to estimate the minimum effective volume of bupivacaine 0.5% resulting in successful block in 50% of patients (MEV50) for ultrasound-guided retroclavicular approach to infraclavicular brachial plexus block.

DETAILED DESCRIPTION:
Two rules were used to stop the study. First stopping rule was a fixed-sample-size. The investigators used an up-and-down method to estimate the threshold for an all-or-none response for present study design. Therefore, for sample size calculation, the investigators applied the formula by Dixon and Massey, n=2(SD/SEM)2 (SD: standard deviation and SEM: standard error of mean). Second stopping rule included demonstration of minimum of five consecutive up-and-down sequences. On the basis of previous studies with similar binary outcomes, the investigators estimated that a priori a minimum of five negative-positive up-and down deflections was required to calculate MEV50.

ELIGIBILITY:
Inclusion Criteria:

* patients who received infraclavicular brachial plexus block for elective elbow, forearm, wrist, or hand surgery
* American Society of Anesthesiologists class I, II or III

Exclusion Criteria:

* patients <18 years old
* >65 years old
* body mass index (BMI) <20 or >35 kg/m2
* inability to provide written informed consent
* refusal of regional anesthesia
* pregnancy
* contraindication for regional anesthesia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults between 18 and 65 years of age with infraclavicular brachial lexus block for elective elbow, forearm, wrist, or hand surgery , were selected in the study.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
The minimum effective volume of bupivacaine 0.5% resulting in successful block in 50% of patients (MEV50) | 30 minutes
  The determination of MEV50 and its 95% confidence interval (CI) was based on the staircase up-and-down method by Dixon and Massey

SECONDARY OUTCOMES:
estimate the minimum effective volume in 95% of patients (MEV95). | 30 minutes
  To calculate the MEV95, data were analyzed using probit transformation and logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Ali Sait Kavakli, M.D., Study Director — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research hospital, Antalya, Turkey (Türkiye)